CLINICAL TRIAL: NCT01777607
Title: The Use of Impella RP Support System in Patients With Right Heart Failure: A Clinical and Probable Benefit Study
Brief Title: The Use of Impella RP Support System in Patients With Right Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Recover Right
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Right Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: IMPELLA® RP

INTERVENTIONS:
Device: IMPELLA® RP

SUMMARY:
The use of Impella RP is safe, feasible and provides a hemodynamic benefit in patients with right ventricular failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have developed signs of right ventricular failure either: A) within 48 hours post-implantation of an FDA approved implantable surgical LVAD (left ventricular assist device )(Cohort A) or B) subsequent to postcardiotomy shock within 48 hours post surgery or post myocardial infarction (Cohort B).
2. Age ≥18 years old
3. Signed Informed consent

Exclusion Criteria

1. INTERMACS 1 patients (Critical cardiogenic shock patient who is "crashing and burning", has life-threatening hypotension and rapidly escalating inotropic or pressor support, with critical organ hypoperfusion often confirmed by worsening acidosis and lactate levels)
2. Evidence of acute neurologic injury
3. RA(right atrium),RV (right Ventricle) and/or PA (pulmonary artery) thrombus
4. Intolerance to anticoagulant or antiplatelet therapies
5. Existing congenital heart disease that would preclude the insertion of the device.
6. Participation in any other clinical investigation that is likely to confound study results or affect study outcome
7. Acute Myocardial Infarction (AMI) with mechanical complications ( ventricular septal defect, myocardial rupture, papillary muscle rupture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Primary Benefit Endpoint | 30 Days
  Survival at 30 days or hospital discharge whichever is longer post device explant or to the next therapy, including transplant, bridge to transplant or destination therapy with FDA approved surgical VAD (Ventricular Assit Device).

CONTACTS AND LOCATIONS:
Overall Officials: William O.Neill, MD, Principal Investigator — Henry Ford Hospital; Mark Anderson, MD, Principal Investigator — Albert Einstein Medical Center
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Anderson MB, Goldstein J, Milano C, Morris LD, Kormos RL, Bhama J, Kapur NK, Bansal A, Garcia J, Baker JN, Silvestry S, Holman WL, Douglas PS, O'Neill W. Benefits of a novel percutaneous ventricular assist device for right heart failure: The prospective RECOVER RIGHT study of the Impella RP device. J Heart Lung Transplant. 2015 Dec;34(12):1549-60. doi: 10.1016/j.healun.2015.08.018. Epub 2015 Sep 8. PMID 26681124